CLINICAL TRIAL: NCT06281223
Title: Study of Brain-spinal Cord Neural Connectivity in Spasticity
Acronym: MOVE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JBR_2023_9
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Spasticity, Muscle
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intraoperative neuroelectrophysiological monitoring — The procedure involves intraoperative neuroelectrophysiological monitoring. The aim is to record the electrical activity of the central and peripheral nervous system at several levels during a neurosurgical procedure.
  The equipment used comes from INOMED and consists of :
  * a recording station (ISIS)
  * scalp corkscrew electrodes (2 to 4 electrodes)
  * a 4-pin FSR spinal cord electrode (Ad-Tech)
  * hook electrodes for roots/radicles (X2)
  * needle electrodes for muscles (X18)
  Electrode placement and recording take place in the operating room while the patient is under general anaesthetic (intubated and sedated).

SUMMARY:
Little is known about the peripheral and central mechanisms of action of selective dorsal rhizotomy surgery for the treatment of spasticity. A better understanding of these mechanisms will enable us to improve the surgical procedure. This will require cortico-medullo-radiculo-muscular recordings never before performed and published in the literature, and the identification of variations in connectivity correlated with the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 to 17 years included
* scheduled for selective rhizotomy surgery
* Having received informed consent to participate in the study (written consent from both parents)
* Affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Contraindications to selective rhizotomy
* History of epilepsy
* Known neurological and/or psychiatric disorders with past and/or current medical treatment, or drug addiction
* Patient under legal protection
* Pregnant or breast-feeding women

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with a diagnosis of spasticity requiring selective rhizotomy in neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
variation in "spontaneous/resting" cortico-medullo-radiculo-muscular synchronization before and after selective rhizotomy surgery | Day 0
  variation in the mean spectral power of the neuronal signal between the brain, spinal cord, roots/radicles and muscles (simultaneous recording levels) before and after surgery.
  Recordings are expressed as currents, themselves defined by waves. Calculating the average spectral power of the neuronal signal at several points is equivalent to quantifying the power of similarity (frequency and amplitude) between two waves.

CONTACTS AND LOCATIONS:
Overall Officials: Pia VAYSSIERE, MD, Study Director — HFAR
Locations (2):
- France (2):
  - Hpu Lenval, Nice
  - HFAR, Paris

IPD SHARING:
Plan to Share IPD: No